CLINICAL TRIAL: NCT07089589
Title: Preoperative Statin Use and Major Adverse Cardiovascular Events in Liver Transplant Recipients: A Multicenter Retrospective Cohort Study
Brief Title: Preoperative Statin Use and Major Adverse Cardiovascular Events in Liver Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Samsung Medical Center (Other); Inje University Haeundae Paik Hospital (Other)
Responsible Party: Principal Investigator, Jun-Gol Song, Professor, Asan Medical Center
Other Study IDs: 2025-0645
Record Dates: First submitted 2025-07-18; First posted 2025-07-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Major Adverse Cardiovascular Events; Liver Transplantation
Keywords: statin; liver transplantation; major adverse cardiovascular events
MeSH Terms: interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Patients who did not receive preoperative statin therapy
- Statin group: Patients who received preoperative statin therapy
  Interventions: Drug: Preoperative Statin Use

INTERVENTIONS:
Drug: Preoperative Statin Use — Administration of any statin medication prior to liver transplantation. Statin therapy was previously prescribed by the treating physician before the transplant procedure, not assigned by the study protocol.
  Other Names: HMG-CoA Reductase Inhibitor
  Groups: Statin group

SUMMARY:
The goal of this multicenter observational study is to determine whether preoperative statin use reduces major adverse cardiovascular events or other complications after liver transplantation. The main question it aims to answer is:

Does preoperative statin use reduce major adverse cardiovascular events or other complications after liver transplantation? The records of participants who already took statins before liver transplantation will be reviewed.

DETAILED DESCRIPTION:
Cardiovascular complications have emerged as a leading cause of early postoperative death following liver transplantation (LT), accounting for over 40% of early deaths. As a result, preventing postoperative cardiac complications has become a critical concern in the management of LT recipients.

Statin therapy has been suggested to improve perioperative and long-term outcomes in various surgical populations, primarily through LDL cholesterol reduction as well as pleiotropic effects, such as enhanced endothelial function and anti-inflammatory actions. However, evidence specifically examining the impact of preoperative statin therapy on cardiovascular outcomes after LT remains limited, highlighting the need for further research in this population.

This study aimed to address the current knowledge gap by investigating the association between preoperative statin use and the incidence of major adverse cardiovascular events within 30 days after liver transplantation in liver transplant recipients. Secondary outcomes included overall mortality, early allograft dysfunction, acute kidney injury, length of stay in the intensive care unit, duration of mechanical ventilation, and myocardial injury after non-cardiac surgery within 3 and 30 days after transplantation.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients aged ≥18 years who underwent liver transplantation

Exclusion Criteria:

* Patients who underwent liver re-transplantation
* Patients with preoperative acute-on-chronic liver failure (ACLF)
* Patients with preoperative fulminant hepatic failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) who underwent liver transplantation at Asan Medical Center, Samsung Medical Center, and Inje University Haeundae Paik Hospital in Korea between January 2008 and January 2026.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2008-01-02 (Actual); Primary Completion 2026-01-25 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
30-day Major Adverse Cardiovascular Events | 30 days after liver transplantation
  The composite of cardiovascular death, heart failure, myocardial infarction, atrial fibrillation, ventricular arrhythmia, ischemic electrocardiogram changes (ST-segment depression or elevation) with chest tightness, pulmonary embolism, and stroke

SECONDARY OUTCOMES:
Overall Mortality | From the date of liver transplantation to May 19, 2025
  Death from any cause after liver transplantation
Acute Kidney Injury | Within 7 days after liver transplantation
  Occurrence of acute kidney injury within 7 days post-transplantation, diagnosed according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria
Early Allograft Dysfunction | Within 7 days after liver transplantation
  Defined as serum bilirubin >10 mg/dL or international normalized ratio (INR) >1.6 on postoperative day (POD) 7, or alanine/aspartate aminotransferases >2000 IU/L within 7 days after transplantation
Intensive Care Unit Length of Stay | From the date of liver transplantation until intensive care unit discharge, up to 600 days
  Total duration (days) of intensive care unit stay after liver transplantation
Mechanical Ventilation Duration | From the date of transplantation until discontinuation of mechanical ventilation, up to 600 days
  Duration (days) of postoperative mechanical ventilation following liver transplantation
Myocardial Injury after Non-Cardiac Surgery (MINS) | Within 3 days and 30 days after liver transplantation
  The incidence of MINS within 3 and 30 days. Defined as a postoperative cardiac TnI level above 40 pg/mL before November 2021, and above 60 pg/mL thereafter, based on the 99th percentile upper reference limit for high-sensitivity TnI assays established in the Korean population

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No